CLINICAL TRIAL: NCT07002008
Title: The Effects of Scapular Stabilization Exercises on Shooting Accuracy and Upper Extremity Performance in Traditional Archery Athletes: A Randomized Controlled Trial
Brief Title: The Effects of Scapular Stabilization Exercises in Traditional Archery Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: archery
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Athletes; Exercise; Archery
Keywords: traditional archery; scapular stabilization; shooting performance; strength; balance; endurance; proprioception
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel assignment interventional model in which participants are randomly allocated into two distinct groups: an intervention group receiving scapular stabilization exercises and a control group continuing with standard archery training. Each participant remains in their assigned group throughout the 8-week intervention period.
  The intervention will be supervised by a physiotherapist aware of group allocation, while pre- and post-intervention measurements will be conducted by evaluators who remain blinded throughout the study. The model is designed to ensure comparability between groups and to assess the specific contribution of scapular stabilization exercises on the targeted outcomes.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Stabilization Exercise Program (Experimental): Frequency: 3 times/week for 8 weeks
  Duration: ~40 minutes per session
  Exercises: Scapular retraction, push-up with plus, scapular depression with resistance band, dipping, forward lean on therapy ball
  Load progression based on 20-rep max tests every 2 weeks
  Conducted under physiotherapist supervision
  Interventions: Other: Scapular Stabilization Exercise
- Control Group (No Intervention): Regular archery training without additional exercises

INTERVENTIONS:
Other: Scapular Stabilization Exercise — Intervention Description:
  The intervention consists of a structured, physiotherapist-supervised scapular stabilization exercise program developed specifically for athletes engaged in traditional archery. The program is designed to enhance scapular alignment, motor control, and dynamic stability by targeting key stabilizing muscles such as the serratus anterior and lower trapezius.
  Participants in the intervention group will continue their standard traditional archery training and will additionally perform the scapular stabilization protocol three times per week for 8 consecutive weeks, with each session lasting approximately 40 minutes.
  The exercise regimen includes:
  Scapular Retraction Exercise (prone position with arm elevation)
  Push-Up Plus Exercise (with scapular protraction emphasis)
  Scapular Retraction and Depression with Elastic Band Resistance
  Dipping Exercise (shoulder elevation and scapular control in seated position)
  Forward Lean Exercise on Therapy Ball (scapular pro
  Arms: Scapular Stabilization Exercise Program

SUMMARY:
This randomized controlled trial aims to investigate the effects of an 8-week scapular stabilization exercise program on shooting accuracy and upper extremity performance in athletes engaged in traditional archery. Thirty licensed archers aged between 15 and 35, with at least 2 years of experience, will be randomly assigned to an intervention group or a control group. The intervention group will receive scapular stabilization exercises in addition to their regular training, while the control group will continue their usual training routine. Pre- and post-intervention evaluations will assess upper extremity strength, stability, proprioception, and shooting performance.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial designed to investigate the effectiveness of scapular stabilization exercises on shooting performance and upper extremity functional capacity in athletes engaged in traditional archery. Traditional archery is a sport that places significant demands on shoulder girdle stability, particularly during the aiming and release phases. Improper scapular positioning and muscular imbalances may negatively impact accuracy and increase the risk of shoulder injuries over time.

Participants will be stratified by age and gender and randomly allocated into two groups: an intervention group performing a standardized scapular stabilization program in addition to regular training, and a control group continuing with regular training alone. The exercise program targets key scapular stabilizers, including the serratus anterior and lower trapezius, with the goal of improving scapular alignment, motor control, and muscular endurance. Exercise progression will be tailored to individual response and load tolerance.

Assessments will include validated performance and functional tests to evaluate changes in upper extremity strength, endurance, proprioception, and shooting accuracy. Pre- and post-intervention assessments will be conducted by blinded evaluators to minimize measurement bias. The study protocol has been designed to ensure methodological rigor, with strict adherence to randomization, blinding, and standardized testing procedures.

This research aims to fill a gap in the literature concerning shoulder health and performance in traditional archery athletes and may provide valuable guidance for clinicians and coaches involved in the training and rehabilitation of overhead sport athletes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 35 years

Licensed traditional archers with at least 2 years of experience

Regular participation in training programs

Willingness to participate and provide informed consent

Exclusion Criteria:

* History of upper extremity orthopedic surgery in the past year

Existing musculoskeletal disorders in the upper extremity

Presence of any neurological disease

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Archery Shooting Performance Score | Baseline and 8 weeks after intervention
  Shooting accuracy will be assessed using a standardized Archery Shooting Score Test. Athletes will perform ten shots at a distance of 18 meters using a standard indoor target with concentric colored scoring rings. The first 4 shots are considered warm-up, and the total score of the final 6 shots will be recorded. Scoring will be based on World Archery guidelines.
Closed Kinetic Chain Upper Extremity Stability Test | Baseline and 8 weeks after intervention
  Upper extremity stability and strength will be evaluated using the Closed Kinetic Chain Upper Extremity Stability Test. Participants will perform hand touches across a 91.4 cm distance while maintaining a modified push-up position. Each trial will last 15 seconds, and the number of touches will be counted. The test will be repeated three times, with 45-second rest intervals, and the average number of touches will be recorded as the final score.
Upper Quarter Y Balance Test | Baseline and 8 weeks after intervention
  Assesses shoulder mobility, proprioception, and balance in three directions (medial, superolateral, inferolateral). The average normalized reach distance (in cm) across three attempts in each direction will be recorded and used to calculate a composite score.
Seated Medicine Ball Throw Test | Baseline and 8 weeks after intervention
  Measures upper extremity explosive power by calculating the average distance (in cm) a 2 kg medicine ball is thrown while seated against a wall with back and head contact maintained. The best 3 of 4 trials will be averaged.
Isometric Upper Extremity Muscle Strength | Baseline and 8 weeks after intervention
  Strength will be assessed using a digital handheld dynamometer. Measurements will be taken in multiple directions including shoulder flexion, extension, abduction, internal and external rotation; elbow flexion and extension; and wrist extension. A maximum of three trials will be performed for each direction, and the highest value will be recorded in Newtons.
Upper Extremity Proprioception | Baseline and 8 weeks after intervention
  Proprioception will be assessed using a digital inclinometer. Participants will be asked to reproduce 90° of shoulder flexion and abduction with their eyes closed. The angular deviation from the target position will be recorded. Lower deviation values will indicate better proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Atıcılar Archery Facility, Bursa Metropolitan Municipality, Bursa, Osmangazi̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Şimşek, D., A. Cerrah, H. Ertan, and M. Tekce. 2013. "The Assessment of Postural Control Mechanisms in Three Archery Disciplines: A Preliminary Study." Pamukkale Journal of Sport Sciences 4 (3): 18-28.
- [Background] Cerrah AO, Simsek D, Soylu AR, Nunome H, Ertan H. Developmental differences of kinematic and muscular activation patterns in instep soccer kick. Sports Biomech. 2024 Jan;23(1):28-43. doi: 10.1080/14763141.2020.1815827. Epub 2020 Sep 15. PMID 32930059